CLINICAL TRIAL: NCT03626311
Title: A Double-Blind, Placebo-Controlled Randomized, Multicenter Study to Assess Changes in Omega-3 Index in Erythrocytes and Health Benefit After 24 Weeks of Daily Consumption of AKBM-3031 (Omega-3 Phospholipids From Krill), Followed by a 24 Week Open-Label Extension, in Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: Omega-3 Replacement With Krill Oil in Disease Management of SLE
Acronym: ORKIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aker BioMarine Human Ingredients AS (Industry)
Collaborators: Ampel BioSolutions, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AMP-004
Record Dates: First submitted 2018-06-06; First posted 2018-08-13 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Lupus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized (1:1) to receive either AKBM-3031 or placebo during the randomized period.The randomized subjects will take (4)1 gram capsules of product or placebo every day, (2) 1 gram capsules in the morning and (2) 1 gram capsules in the evening, for a total of 4 grams per day for the first 24 weeks (randomized period). All subjects may continue to a 24-week extension (Open Label Extension) of open-label AKBM-3031, 4 grams/day. The total study duration per subject is 48 weeks. With about 4 months for site activation and 12 months for enrollment, the entire study is expected to complete in approximately 116 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AKBM-3031 (Experimental): 4g/day (2 capsules BID)
  Interventions: Dietary Supplement: AKBM-3031
- Placebo (Placebo Comparator): 4g/day (2 capsules BID)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: AKBM-3031 — Krill are shrimp-like small crustaceans (up to 6 cm) found in all the world's oceans, but mostly in the Arctic and Antarctic polar seas. Krill are rich in the long-chain omega-3 polyunsaturated fatty acids or LC-PUFAs eicosapentaenoic acid (EPA, C20:5n3) and docosahexaenoic acid (DHA, C22:6n3). The lipid pool of krill is composed of phospholipids and triglycerides and the LC-PUFAs are primarily in the phospholipid fraction.
  The product is produced under food Good Manufacturing Practice (GMP) regulations and has status as GRAS or Generally Recognized As Safe. GRAS is defined by the US Food and Drug Administration (FDA) as a substance that is generally recognized, among qualified experts, to be safe under the conditions of its intended use.
  Other Names: Krill Oil
  Arms: AKBM-3031
Other: Placebo — The placebo will be provided in capsules looking exactly as the krill oil capsules and will contain a fatty acid mixture (olive oil, corn oil, palm oil and medium chain triglycerides) which has the same composition as the average European diet (26.0% C16:0, 4.6% C18:0, 35.8% C18:1n9, 16.7% C18:2n6, 2.1% C18:3n3, 0% C20:4n6 and 14.8% other compounds) and contains no EPA or DHA.
  Arms: Placebo

SUMMARY:
A randomized, double-blind controlled, multicenter study in SLE patients given AKBM-3031or placebo for 24 weeks (randomized period) and followed by an open label extension (OLE) treatment with AKBM-3031 for the next 24 weeks. Patients will be maintained on stable doses of background medications, except for glucocorticoids. Decreases in doses of glucocorticoids will be encouraged during the first 20 weeks of both the randomized and open label extension portions of the trial. Stable doses of glucocorticoids and other background medications are required during weeks 20-22 and 44-48.If indicated by the PI, brief increases in corticosteroids are permitted during the first 20 weeks of both the blinded and open label extension portion of the trial. The increase in prednisone (or equivalent) dose is limited to 2X the back-ground level to a maximum of20 mg/day for a maximum of 1 week (7 days) or to a single administration of intravenous methylprednisolone or equivalent at a maximum dose of 500mg. Stable doses of glucocorticoids and other background medications are required during weeks 20-22 and 44-48

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged at least 18 years old.
2. Capable of giving written consent on an Institutional Review Board or IRB-approved Informed Consent Form prior to any study-specific evaluation
3. Have a clinical diagnosis of SLE with at least 4 of the 11 American College of Rheumatology (ACR) criteria as modified in 1997 or meeting SLICC criteria
4. SLE activity (SLEDAI ≥6)
5. On a stable SLE treatment regimen consisting of a stable dosage of any of the following medications for a period of at least 30 days prior to Baseline (i.e., day of 1st dose of study agent):

   1. Corticosteroids. Corticosteroids (< 20 mg prednisone or equivalent per day)
   2. Hydroxychloroquine or equivalent anti-malarial
   3. Other immunosuppressive or immunomodulatory agents including methotrexate, azathioprine, leflunomide, mycophenolate (including mycophenolate mofetil, mycophenolate mofetil hydrochloride, and mycophenolate sodium at no more than 2 grams/day), calcineurin inhibitors (e.g., tacrolimus,cyclosporine)
   4. Belimumab dose must be stable for 60 days prior to Baseline
   5. Cyclophosphamide dose must be stable for the last 90 days prior to Baseline
   6. Have not received rituximab within 6 months
6. Have a low habitual consumption of fatty fish and seafood, defined as a frequency of twice per month or less; see Addendum 1 for a list of fish and seafood considered to be fatty.

Exclusion Criteria:

Patients are excluded from the study if any of the following criteria are met:

1. Have rapidly progressive neurologic or renal disease
2. Currently taking an omega-3 prescription drug (e.g. Lovaza®, Vascepa®, etc.) or as medical food (e.g. Vascazen®, Vayarin, Onemia™etc.)
3. Present or recent use (within 3 months of screening) of any OTC fish or krill oil dietary supplement., or any long-chain omega-3 fatty acid dietary supplement (e.g.,MegaRed)
4. Have severe lupus kidney disease (defined by proteinuria > 6 gm/24 hour or equivalent using spot urine protein to creatinine ratio, or serum creatinine > 2.5mg/dL)
5. Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases not related to SLE (i.e., diabetes, cardiovascular, pulmonary, hematologic, gastrointestinal, neurological, or infectious) which, in the opinion of the treating physician, could confound the results of the study or put the patients at undue risk
6. Have received intravenous glucocorticoids at a dosage of ≥ 500 mg daily within the past month
7. Require anti-coagulation with coumadin, clopidogrel, dalteparin, dypyridamole, enoxaparin, heparin or ticlopidine. Low dose aspirin (<325 mg/day) is permitted.
8. Receiving orlistat (Xenical, Alli) and have refused to discontinue at baseline and throughout the trial.
9. History of allergy to seafood or shellfish
10. Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 364 days prior to Baseline
11. Are pregnant or lactating
12. Recent participation in a clinical trial with an experimental agent in the past 6 weeks, or 5 half-lives of the study drug, whichever is longer
13. Have a Grade 3 or greater laboratory abnormality based on the Adverse Event Severity Grading Tables (CTCAE), except for the following that are allowed:

    1. Stable Grade 3 partial thromboplastin time (PTT) due to lupus anticoagulant and not related to liver disease or anti-coagulant therapy
    2. Stable Grade 3 hypoalbuminemia due to chronic lupus nephritis, and not related to liver disease
    3. Stable Grade 3 gamma glutamyl transferase (GGT) elevation due to lupus hepatitis, and not related to alcoholic liver disease, uncontrolled diabetes, or viral hepatitis. If present, any abnormalities in the ALT or Alanine Transaminase and/or AST or Aspartate Transaminase must be < Grade 2.
    4. Stable Grade 3 neutropenia or stable Grade 3 white blood cell count due to lupus.
14. Patients will be excluded from the study based on the following bone marrow, hepatic and renal function values:

    1. Hemoglobin: < 8.0 gm/dL
    2. Platelets: <50,000/mm
    3. ANC < 1.0 x 103/mm
    4. AST or ALT >2.5 x Upper Limit of Normal unless related to primary disease.
    5. Creatinine clearance ≤ 25ml/min per 1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2021-08-21 (Actual); Study Completion 2021-08-21 (Actual)

PRIMARY OUTCOMES:
Difference in the ratio of omega-3 to omega-6 measured through lab tests on red blood cells from baseline through the end of the study in patients with generalized lupus. | Baseline to 24 weeks

SECONDARY OUTCOMES:
Effect of correction of omega-3 deficiency measured by SLE biomarkers of immune function. | Baseline to 24 weeks
Effect of correction of omega-3 deficiency measured by both clinician and patient reported outcomes collected at clinic visits. | Baseline to 24 weeks
Change in health related quality of life measured using the Medical Outcomes study Short Form 36 (SF-36). | Baseline to 24 weeks
  Both physical component scores (PCS) and mental component scores (MCS) will be assessed. Change in both PCS and MCS will be evaluated over the time of this study. The SF-36 is a patient recorded survey of health related quality of life, consisting of the evaluation of 8 domains, and then scored from 0-100. The higher score correlates to better health-related quality of life. The mean for healthy individuals is 50.
Difference of number of patients with reported adverse events or changes in lab parameters while taking AKBM-3031. | Baseline to 24 weeks
  Examples of patient reported adverse events include gastrointestinal symptoms, infection, unexplained bleeding, etc. Examples of lab parameters indicating an adverse event are changes in liver function tests, urinalysis, and hematologic parameters (which could be considered an adverse event).

CONTACTS AND LOCATIONS:
Locations (19):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Wallace Rheumatic Studies Center, LLC, Beverly Hills, California
  - UC Irvine Health, Orange, California
  - University of Miami, Miami, Florida
  - Rush Medical Center, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Northwell Health, Great Neck, New York
  - Feinstein Institute for Medical Research, Manhasset, New York
  - Hospital for Special Surgery, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
- Canada (4):
  - Lupus Clinic-Mary Pack Arthritis Centre, Vancouver, British Columbia
  - McMaster University Medical Center, Hamilton, Ontario
  - McGill University Health Centre-The Montreal General Hospital, Montreal, Quebec
  - University of Laval, Québec

REFERENCES:
- [Derived] Salmon J, Wallace DJ, Rus V, Cox A, Dykas C, Williams B, Ding Y, Hals PA, Johnsen L, Lipsky PE. Correction of omega-3 fatty acid deficiency and improvement in disease activity in patients with systemic lupus erythematosus treated with krill oil concentrate: a multicentre, randomised, double-blind, placebo-controlled trial. Lupus Sci Med. 2024 Jul 14;11(2):e001201. doi: 10.1136/lupus-2024-001201. PMID 39009356